CLINICAL TRIAL: NCT07071194
Title: The Effect of Osteopathic Manipulative Treatment on Respiratory Function in Patients With Asthma
Brief Title: Asthma and Osteopathic Manipulative Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Nancy Wasserbauer-Kingston, Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20250241
Record Dates: First submitted 2025-06-19; First posted 2025-07-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Osteopathic Manipulative Treatment; Lung inflammation; Improved breathing
MeSH Terms: conditions — Asthma; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group using OMT (Experimental): Patients in the treatment group will undergo OMT using sub-occipital release, rib raising, doming the diaphragm, thoracic inlet release and myofascial techniques.
  Interventions: Procedure: OMT
- Control group (Active Comparator): Patients in the control group will undergo light touch in similar locations to above performed OMT.
  Interventions: Other: Light touch

INTERVENTIONS:
Procedure: OMT — Patients in the treatment group will undergo OMT using sub-occipital release, rib raising, doming the diaphragm, thoracic inlet release and myofascial techniques.
  Arms: Treatment group using OMT
Other: Light touch — Patients in the control group will undergo light touch in similar locations to OMT.
  Arms: Control group

SUMMARY:
Asthma is a common respiratory condition that can be difficult to control despite the use of medications such as inhalers, oral steroids or even injectable medications. Osteopathic Manipulative Treatment (OMT) is a hands-on technique used to improve the chest structure and function and may help in improving breathing. Previous research showed that OMT in asthma patients, can improve the movement of the ribs and improve the "peak flow" which is the maximum rate at which a person can exhale air after taking a deep breath. However, no studies have evaluated the impact of OMT on lung inflammation.

This single-site research study at University Hospitals aims to evaluate whether Osteopathic Manipulative Treatment (OMT) can reduce lung inflammation and improve breathing and lung function in adult patients with asthma. The lung function will be evaluated by Spirometry which is a test that measures how much air you can breathe in and out of your lungs, as well as how quickly and easily you can exhale air. The lung inflammation will be measured using a device that can detect how much you are breathing out Nitric Oxide which is a gas produced by inflamed cells in the lungs, this test is called: Fractional exhaled Nitric Oxide or FeNO. Approximately 100 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients in Allergy and Immunology Associates clinic diagnosed with asthma ages 18-60 years old with an elevated FENO

Exclusion Criteria:

* Use of oral steroids within the last 4 weeks
* Use of biologic medications
* Diagnosis of pregnancy, osteoporosis, congestive heart failure, renal failure, cirrhosis, or cancer
* Inability to lay recumbent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fractionated Exhaled Nitric Oxide (FeNO) values as measured by NIOX FeNO device | Baseline, after OMT treatment (up to 30 minutes), day 10
Change in Peak Expiratory Flow values as measured by EasyOne Air Spirometer device | Baseline, after OMT treatment (up to 30 minutes), day 10

SECONDARY OUTCOMES:
Change in Ease of breathing as measured by Post-OMT Questionnaire | Baseline and day 10
  The post_OMT Questionnaire scores ease of breathing on a Likert scale of 1-0 with 1 being difficult to breathe and 10 being easy to breath
Change in Rib Cage mobility as measured by Post-OMT Questionnaire | Baseline and day 10
  The post_OMT Questionnaire scores Rib Cage mobility on a Likert scale of 1-0 with 1 being stiff and 10 being mobile
Change in chest tightness as measured by Post-OMT Questionnaire | Baseline and day 10
  The post_OMT Questionnaire scores chest tightness on a Likert scale of 1-0 with 1 being tight and 10 being loose

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wasserbauer-Kingston, DO, Principal Investigator — University Hospitals
Locations (1):
- Allergy Immunology Associates, Mayfield Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No